CLINICAL TRIAL: NCT00555919
Title: Randomized Phase II Study to Investigate the Efficacy, Safety and Tolerability of ZK 230211 (25 mg vs. 100 mg) as Second-line Endocrine Therapy for Postmenopausal Women With Hormone Receptor-positive Metastatic Breast Cancer
Brief Title: ZK 230211 in Postmenopausal Woman With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91484; 2005-005581-36 (EudraCT Number); 309821 (Other: Company internal)
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer stage IV; Metastatic breast cancer; mBC; Stage IV breast cancer; Hormone receptor positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — lonaprisan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Lonaprisan (ZK 230211, BAY86-5044)
- Arm 2 (Experimental)
  Interventions: Drug: Lonaprisan (ZK 230211, BAY86-5044)

INTERVENTIONS:
Drug: Lonaprisan (ZK 230211, BAY86-5044) — 25 mg daily oral treatment
  Arms: Arm 1
Drug: Lonaprisan (ZK 230211, BAY86-5044) — 100 mg daily oral treatment
  Arms: Arm 2

SUMMARY:
Randomized phase II study to investigate the efficacy, safety and tolerability of ZK 230211 (100 mg vs. 25 mg) as second-line endocrine therapy for postmenopausal women with hormone receptor-positive metastatic breast cancer.Once the cancer has spread beyond the lymph nodes to areas such as e.g. the skin, soft tissues, lung, and liver it is called metastatic breast cancer. Patients who have been diagnosed with metastatic breast cancer that has progressed since their previous cancer treatment and that cannot be removed completely by surgery are eligible to be treated within this trial.Treatment with a new drug called Progesterone Receptor Antagonist ZK 230211 (ZK PRA) targets the progesterone receptor which may be expressed on breast cancer tumour cells. Therefore only patients with this progesterone receptor on their tumour cells can be included in this study.Progesterone receptor antagonists (including onapristone) have already shown efficacy in postmenopausal women with advanced breast cancer (Klijn et al. 2000). This phase II study investigates the efficacy (proof of concept), safety and tolerability of ZK PRA at two dose levels (25 mg and 100 mg) before initiating pivotal phase III trials.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women defined as: aged >/= 50 years with amenorrhea for at least 12 months or aged < 50 years with 6 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) level within postmenopausal range (> 40 mIU/ml) or having undergone bilateral oophorectomy
* Histologically or cytologically confirmed breast cancer
* Metastatic breast cancer (Stage IV according to UICC - Union Internationale Contre Cancer - criteria, Version 6)
* Progesterone receptor-positive tumors
* Patients must be considered candidates for endocrine therapy (no other therapies for breast cancer are required)
* Disease progression after first-line endocrine therapy for advanced breast cancer (i.e. with tumor remission or stabilization lasting at least 3 months under endocrine therapy)
* At least one measurable or non-measurable tumor lesion (according to RECIST criteria)
* WHO Performance status 1
* Adequate function of major organs and systems:

  * Hematopoietic:

    * Hemoglobin: 10 g/dL
    * Absolute neutrophil count: 1,500/mm3
    * Platelet count: 100,000/mm3
  * Hepatic:

    * Total bilirubin: 1.5 times the upper limit of normal
    * AST/ALT: 2.5 times the upper limit of normal
  * Renal: Creatinine: 1.5 times the upper limit of normal
  * Gynecological: Endometrial thickness (in non-hysterectomized women) </= 10 mm double layer
  * No other uncontrolled concurrent illness
* Adequate recovery from previous surgery, radiation and chemotherapy
* Written informed consent

Exclusion Criteria:

* Presence of any of the following conditions:

  * life-threatening metastatic visceral disease (extensive hepatic involvement)
  * any metastases to the central nervous system (CNS)
  * pulmonary lymphangitic metastases involving more than 50% of the lung
* More than one prior endocrine treatment for advanced breast cancer
* Previous combination of endocrine treatment with any other type of treatment (except chemotherapy), or previous sequential endocrine treatments (if there was disease progression between treatments) are not permitted in this trial.
* Patients with breast cancer HER-2 positive or with unknown HER-2 status are not eligible.
* Malignancies or history of prior malignancy other than carcinoma in situ of the cervix or uterus, or basal and squamous cell carcinoma of the skin
* Intake of CYP3A4 inhibitors less than 2 weeks before start of study treatment
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds (ms)
* A history of additional risk factors for TdP (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* The use of concomitant medications that prolong the QT/QTc interval
* Other investigational drug therapies less than 4 weeks or at least 5 half-lives before start of study treatment (less than 4 weeks for faslodex and less than 2 weeks for any other endocrine therapy)
* Expectation that the patient will not be able to complete at least 3 months of therapy
* Unwillingness or inability to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-03; Primary Completion 2010-04 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy (clinical benefit) of two doses of ZK PRA (25 mg and 100 mg) when administered once daily p.o. | month 3, month 6

SECONDARY OUTCOMES:
To evaluate safety and tolerability | ongoing thoughout the trial
To evaluate the pharmacokinetics of ZK PRA | baseline, month1,2,6
To evaluate the effect of ZK PRA on quality of life (QoL) | baseline, month 1,2,3,4,5,6
To perform exploratory analysis of biomarkers | baseline, month 1, 3
Progression-free survival (PFS) | end of study
Objective response rate (ORR) / Duration of response - in the subset of patients with measurable disease | end of study
Duration of Clinical Benefit | end of study
Overall Survival (OS) | end of study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (28):
- Austria (4):
  - Salzburg, Salzburg
  - Vienna, Vienna
  - Graz
  - Innsbruck
- Finland (2):
  - Turku
  - Vaasa
- France (6):
  - Lille
  - Lyon
  - Montpellier
  - Nantes
  - Paris
  - Reims
- Germany (5):
  - Tübingen, Baden-Wurttemberg
  - Erlangen, Bavaria
  - Frankfurt am Main, Hesse
  - Rostock, Mecklenburg-Vorpommern
  - Kiel, Schleswig-Holstein
- Rozzano, Milano, Italy
- Poland (4):
  - Bialystok
  - Gdansk
  - Olsztyn
  - Poznan
- Madrid, Madrid, Spain
- Sweden (3):
  - Gothenburg
  - Sundsvall
  - Vaxjo
- Sankt Gallen, Canton of St. Gallen, Switzerland
- Nottingham, United Kingdom

REFERENCES:
- [Background] Jonat W, Bachelot T, Ruhstaller T, Kuss I, Reimann U, Robertson JFR. Randomized phase II study of lonaprisan as second-line therapy for progesterone receptor-positive breast cancer. Ann Oncol. 2013 Oct;24(10):2543-2548. doi: 10.1093/annonc/mdt216. Epub 2013 Jun 20. PMID 23788750